CLINICAL TRIAL: NCT02080624
Title: Phase II, Randomized, Triple Blind, Intra-individually Placebo-controlled Clinical Trial to Assess the Efficacy and Safety of Topical Rapamycin Associated With Pulsed Dye Laser in Patients With Sturge-Weber Syndrome.
Brief Title: Efficacy and Safety Study of Topical Rapamycin Associated With Pulsed Dye Laser in Patients With Sturge-Weber Syndrome
Acronym: RSW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple
Other Study IDs: RSW2011; 2010-024078-20 (EudraCT Number)
Record Dates: First submitted 2013-04-18; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2013-10

CONDITIONS: Sturge- Weber Syndrome
MeSH Terms: conditions — Brain Stem Infarctions | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapamycin (Experimental): Topical rapamycin applied once a day
  Interventions: Drug: Drug: Topical Rapamycin

INTERVENTIONS:
Drug: Drug: Topical Rapamycin — After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study.
  A medical history, which involves questions about your health history, any medications you are taking or plan to take, any allergies and the treatments you received for your CM.
  A physical exam, during which you will be asked about any problems that you might be having. Additionally, your clinician will check your vital signs (blood pressure, heart rate, weight and height). The doctor will also evaluate your performance status, which indicates how much your illness affects your activity level.
  Blood tests, which will be done to make sure your hemogram, triglyceride and cholesterol levels are normal.
  A pregnancy test for females will be done to check that you are not pregnant. If theses tests show that you are eligible to participate in the research study, you will begin the study treatment.
  Other Names: topical rapamycin 1%

SUMMARY:
Sturge-Weber syndrome (SWS) is a rare congenital neuro-cutaneous disorder considered as a rare or orphan disease. SWS is characterized by a capillary vascular malformation (CM) localized on the skin of the face, eyes and central nervous system. Given the localization and the extent of the CM, children with SWS are particularly prone to developing severe psychological problems. The standard treatment for CM is pulsed dye laser (PDL) although in these cases whitening of the lesion is rarely achieved. Combining topical rapamycin, a specific inhibitor of the mammalian target of rapamycin, with PDL is hypothesised to be a good therapeutic option in these patients.

DETAILED DESCRIPTION:
Patients with SWS will be treated with 2 sessions of PDL in the lateral part of the CM separated by an interval of 6 weeks and with 1% topical rapamycin or placebo in the superior or inferior half, both applied once a day for 12 weeks. The clinical response will be analyzed using a morphologic and chromatographic computerised system and with spectrometry. Histological response will be evaluated also. For that purpose, we will make 4 biopsies, one in each quadrant (quadrant treated with PDL and placebo, quadrant treated with PDL and rapamycin, quadrant treated only with rapamycin and quadrant treated only with placebo)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: All patients must have the diagnostic criteria for Sturge-Weber syndrome.
* Age: patients must be greater than 16 years and less than or equal to 21 years of age at the time of study entry.
* Capillary malformation: patients must have CM on the face.
* Investigational drug: Patients must not have received an investigational drug within 3 months.
* Females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the time they are receiving the study drug and for 3 months thereafter. Abstinence is an acceptable method of birth control. Women of childbearing potential will be given a pregnancy test prior to administration of rapamycin and must have a negative pregnancy test.
* Intellectual capacity to understand the information given and able to comply with the protocol and safety monitoring requirements of the study in the opinion of the investigator.
* Signed informed consent/assent.

Exclusion Criteria:

* Patients with diagnosis of Sturge-Weber syndrome without facial CM.
* Patients with another cutaneous disease on the CM area.
* Patients that will be applying another topical cream on the CM area.
* Chronic treatment with systemic steroids or another immunosuppressive agent. Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Patients who:

  * have had a major surgery or significant traumatic injury within 2 weeks of start of study drug;
  * have not recovered from the side effects of any major surgery (defined as requiring general anesthesia but excluding a procedure for insertion of central venous access), or
  * may require major surgery during the course of the study.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * symptomatic congestive heart failure of New York heart Association Class III or IV.
  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
  * severely impaired lung function.
  * uncontrolled diabetes as defined by fasting serum glucose greater than 1.5 upper limit of normal.
  * active (acute or chronic) or uncontrolled severe infections.
  * liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
* A known history of HIV seropositivity or known immunodeficiency.
* Women who are pregnant or breast feeding.
* Patients who have received prior treatment with an inhibitor of mammalian target of rapamycin.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol or who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in morphologic, chromatographic and spectrometric scores at week 6 | Baseline, Week 6
  Change Outcome Measure
Change from baseline in morphologic, chromatographic and spectrometric scores at week 12 | Baseline, Week 12
  Change Outcome Measure
Change from baseline in morphologic, chromatographic and spectrometric scores at week 18 | Baseline, Week 18
  Change Outcome Measure
Histological response at 12 weeks. | 12 weeks
  Efficacy Outcome Measure

SECONDARY OUTCOMES:
Adverse events at baseline | At the beginning of the intervention
Adverse events at 6 weeks | 6 weeks after the beginning of the intervention
Adverse events at 12 weeks | 12 weeks after the beginning of the intervention
Adverse events at 18 weeks | 18 weeks after the beginning of the intervention
Total blood cholesterol level (mg/dL) at baseline. | At the beginning of the intervention
Total blood cholesterol level (mg/dL) at 6 weeks. | 6 weeks after the beginning of the intervention
Blood concentration of triglycerides (mg/dL) at baseline. | At the beginning of the intervention
Blood concentration of triglycerides (mg/dL) at 6 weeks. | At 6 weeks after the beginning of the intervention
Blood concentration of hemoglobin (g/dL) at baseline. | At the beginning of the intervention
Blood concentration of hemoglobin (g/dL) at 6 weeks. | At 6 weeks after the beginning of the intervention
Blood count of leukocytes (number of cells/mL) at baseline. | At the beginning of the intervention.
Blood count of leukocytes (number of cells/mL) at 6 weeks. | At 6 weeks after the beginning of the intervention.
Blood platelet count (number of platelets/mL) at baseline. | At the beginning of the intervention.
Blood concentration of rapamycin (ng/ml) at baseline. | At the beginning of the intervention.
Blood concentration of rapamycin (ng/ml) at 6 weeks. | At 6 weeks after the beginning of the intervention.
Blood platelet count (number of platelets/mL) at 6 weeks. | At 6 weeks after the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maider Pretel, MD PhD, Principal Investigator — Clinica Universidad de Navarra; Leyre Aguado, MD PhD, Principal Investigator — Clinica Universidad de Navarra; Laura Marqués, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain